CLINICAL TRIAL: NCT04169737
Title: A Randomized Phase II Study of Acalabrutinib (ACA) + Venetoclax (VEN) +/- Early Obinutuzumab (OBIN) for Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Acalabrutinib and Venetoclax With or Without Early Obinutuzumab for the Treatment of High Risk, Recurrent, or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0565; NCI-2019-06675 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0565 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (acalabrutinib, venetoclax, obinutuzumab) (Active Comparator): Patients receive acalabrutinib PO BID on days 1-28. Beginning cycle 3, patients receive venetoclax PO BID on days 1-28. Patients who are BM MRD4-positive or in PR also receive obinutuzumab IV over 4-6 hours on days 1, 2, 8, and 15 of cycle 15 and day 1 of cycles 16-20. Treatment repeats every 28 days (or 42 days for cycle 14) for up to 26 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib; Biological: Obinutuzumab; Drug: Venetoclax
- Arm II (acalabrutinib, venetoclax, early obinutuzumab) (Experimental): Patients receive acalabrutinib PO BID on days 1-28 beginning cycle 2 and venetoclax PO BID on days 1-28 beginning cycle 3. Patients also receive obinutuzumab IV over 4-6 hours on days 1, 2, 8, and 15 of cycle 1 and day 1 of cycles 2-6. Patients who are BM MRD4-positive or in PR receive obinutuzumab IV over 4-6 hours on day 1 cycles 15-20. Treatment repeats every 28 days (or 42 days for cycle 14) for up to 26 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib; Biological: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well acalabrutinib and venetoclax with or without early obinutuzumab work for the treatment of chronic lymphocytic leukemia or small lymphocytic lymphoma that is high risk, has come back (recurrent), or does not respond to treatment (refractory). Acalabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Venetoclax may stop the growth cancer cells by blocking BCL-2 protein needed for cell growth. Immunotherapy with monoclonal antibodies, such as obinutuzumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving acalabrutinib and venetoclax together with early obinutuzumab may improve clinical outcomes and control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate improvement in bone marrow (BM) undetectable-minimal residual disease,10-4 sensitivity (MRD4) from 40% to 70% after 7 courses of combined acalabrutinib (ACA) and venetoclax (VEN) (end of C9 overall) with addition of early obinutuzumab (OBIN). (Treatment-naive [TN] cohort) II. Demonstrate improvement in BM undetectable-MRD4 from 40% to 70% after 12 courses of combined acalabrutinib (ACA) and venetoclax (VEN) (end of cycle [C]14 overall) with addition of early obinutuzumab (OBIN). (Relapsed/refractory [R/R] cohort)

SECONDARY AND EXPLORATORY OBJECTIVES:

I. Determine the safety of combined acalabrutinib, venetoclax obinutuzumab. II. Determine the overall best response rates (complete response [CR], partial response [PR], overall response [OR]) for each cohort and each treatment arm by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 criteria.

III. Estimate the time to best response for each cohort and each treatment arm with this combination.

IV. Estimate the progression-free (PFS) for each cohort and each treatment arm. V. Estimate proportion of patients with blood/BM undetectable-MRD4, blood/BM undetectable-MRD6 (10-6 sensitivity), CR after 12 and 24 courses combination with VEN (end of C14 and C26 overall) (by cohort and OBIN status).

VI. Determine the proportion of patients who receive late OBIN (C15-C20 overall) and conversion rate for blood/BM undetectable-MRD4 and blood/BM undetectable-MRD6 and CR in those who receive late OBIN.

VII. Correlate plasma cell-free deoxyribonucleic acid (DNA) (cfDNA) with cell-based blood/BM undetectable-MRD4, blood/BM undetectable-MRD6 status at all response assessment time points.

VIII. Determine proportion of patients who discontinue treatment early based on undetectable-MRD results.

IX. Determine time-to-blood MRD6 relapse for those who achieve undetectable-MRD6.

X. Determine response to re-treatment upon relapse. XI. Assess clonal evolution at relapse and correlate with plasma cell-free DNA (cfDNA).

XII. Determine OBIN pharmacokinetics - free drug level assessments to optimize dosing.

XIII. Determine VEN pharmacokinetics - free drug levels to assess changes in exposure with combination.

XIV. Determine ACA pharmacokinetics - free drug levels to assess changes in exposure with combination.

XV. Identify predictive markers for response and outcomes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28. Beginning cycle 3, patients receive venetoclax PO BID on days 1-28. Patients who are BM MRD4-positive or in PR also receive obinutuzumab intravenously (IV) over 4-6 hours on days 1, 2, 8, and 15 of cycle 15 and day 1 of cycles 16-20. Treatment repeats every 28 days (or 42 days for cycle 14) for up to 26 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive acalabrutinib PO BID on days 1-28 beginning cycle 2 and venetoclax PO BID on days 1-28 beginning cycle 3. Patients also receive obinutuzumab IV over 4-6 hours on days 1, 2, 8, and 15 of cycle 1 and day 1 of cycles 2-6. Patients who are BM MRD4-positive or in PR receive obinutuzumab IV over 4-6 hours on day 1 cycles 15-20. Treatment repeats every 28 days (or 42 days for cycle 14) for up to 26 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of CLL/SLL and indication for treatment by 2018 iwCLL criteria:

   Cohort 1: Untreated patients with at least 1 high-risk feature (del(17p) or mutated TP53 or del(11q) or unmutated IGHV or complex karyotype) OR ≥65 years of age Cohort 2: Relapsed after and/or refractory to at least one prior therapy
2. Age 18 years or older
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2
4. Adequate renal and hepatic function:

   * Total bilirubin ≤1.5 x upper limit of normal (ULN) or ≤3 x ULN for patients with Gilbert's disease
   * Creatinine clearance >50 mL/min (calculated according to institutional standards or using Cockcroft-Gault, MDRD, or CKD-EPI formula)
   * ALT and AST ≤3.0 x ULN, unless clearly due to disease involvement
5. Absolute neutrophil count greater than 750 neutrophils/L, unless thought to be due to marrow infiltration with CLL. Platelet count of greater than 30,000/µl, with no platelet transfusion in 2 weeks prior to registration , unless thought to be due to marrow infiltration with CLL.
6. Women of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (β-hCG) pregnancy test result within 7 days prior to the first dose of study drugs and must agree to use an effective contraception method during the study and for 2 days after the last dose of acalabrutinib, 30 days after the last dose of venetoclax, or 18 months after the last dose of obinutuzumab, whichever is longer. Women of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy. Men who are sexually active must agree to use highly effective forms of contraception with the addition of a barrier method (condom) during the study and for 30 days after the last dose of venetoclax and for 18 months after the last dose obinutuzumab, whichever is longer.
7. Free of prior malignancies for 2 years with exception of patients diagnosed with basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast, who are eligible even if they are currently treated or have been treated and/or diagnosed in the past 2 years prior to study enrolment. If patients have another malignancy that was treated within the last 2 years, such patients may be enrolled, if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at MD Anderson Cancer Center, and after consultation with the Principal Investigator.
8. Patients must provide written informed consent.

Exclusion Criteria:

1. Prior treatment with combined BTKi and BCL2i where patients do not achieve at least partial response or progress and need new treatment within 2 years of completing fixed-duration combined treatment.
2. Major surgery, radiotherapy, chemotherapy, biologic therapy, immunotherapy, investigational therapy or live virus vaccination within 3 weeks prior to the first dose of the study drugs, unless patients have rapidly progressive disease, in which case, washout will be 3 drug half-lives
3. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
4. Uncontrolled clinically significant active infection (viral, bacterial, and fungal)
5. Known positive serology for human immunodeficiency virus (HIV), due to potential drug-drug interactions between anti-retroviral medications and the study drugs
6. Active hepatitis B infection (defined as the presence of detectable HBV DNA, HBe antigen or HBs antigen). Subjects with serologic evidence of prior vaccination (HBsAg negative, anti-HBs antibody positive, anti-HBc antibody negative) are eligible. Patients who are HBsAg negative/HBsAb positive but HBcAb positive are eligible, provided HBV DNA is negative.
7. Active hepatitis C, defined by the detectable hepatitis C RNA in plasma by PCR
8. Active, uncontrolled autoimmune phenomenon (autoimmune hemolytic anemia or immune thrombocytopenia) requiring steroid therapy with >20mg daily of prednisone dose or equivalent
9. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
10. Patient is pregnant or breast-feeding
11. Concurrent use of warfarin
12. Received strong CYP3A inhibitors or strong CYP3A inducers within 7 days of starting study drugs and throughout venetoclax administration
13. Consumed grapefruit, grapefruit products, Seville oranges, or star fruit within 7 days of starting venetoclax
14. Known bleeding disorder or history of stroke or intracranial hemorrhage within past 6 months
15. Malabsorption syndrome or other condition that precludes enteral route of administration
16. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
Disease assessment of bone marrow (BM) undetectable-minimal residual disease,10-4 sensitivity (MRD4) (Treatment-naive [TN] cohort) | Up to 1 year end of cycle 9; each cycle 28 days
Disease assessment of BM undetectable-MRD4 (Relapsed/refractory [R/R] cohort) | Up to 1 year end of cycle 14; each cycle 28 days

SECONDARY OUTCOMES:
Incidence of adverse events | From the start of combination therapy up to end of cycle 4; each cycles 28 days
  Toxicities (defined as prolonged grade >= 3 neutropenia or thrombocytopenia lasting > 42 days; febrile neutropenia; hospitalization due to infection; early death; major bleeding due to thrombocytopenia) will be monitored for each treatment arm separately using the Bayesian method of Thall, Simon and Estey.

CONTACTS AND LOCATIONS:
Overall Officials: William G Wierda, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org